CLINICAL TRIAL: NCT02584049
Title: Effects of Osteopathic Treatment in the Management of Care-induced Pain in Elderly Care, in Follow-up Care and Rehabilitation Geriatric
Brief Title: Osteopathic Medicine in the Management of Care-induced Pain in Elderly Care (OGéDIS)
Acronym: OGéDIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely because of the low inclusion rate (1 inclusion in 16 months), the low patient potential and the difficulty of finding new recruiting centres.
Sponsor: Hôpital NOVO (Other)
Collaborators: ESO Paris Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHRD0215
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Pain
Keywords: Osteopathic treatment; Care-induced Pain; Pain; Elderly
MeSH Terms: conditions — Pain | interventions — Osteopathic Physicians

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathy (Active Comparator): 3 sessions of Osteopathic treatment in addition to the usual follow
  Interventions: Other: Osteopathy
- Sham osteopathy (Sham Comparator): 3 sessions of Sham osteopathy treatment in addition to the usual follow
  Interventions: Other: Sham osteopathy

INTERVENTIONS:
Other: Osteopathy — 3 sessions of osteopathy during 60 minutes each
  Arms: Osteopathy
Other: Sham osteopathy — 3 sessions of sham osteopathy during 60 minutes each
  Arms: Sham osteopathy

SUMMARY:
The purpose of this study is to evaluate effects of Osteopathic Treatment in the Management of Care-induced pain in Elderly care, in Follow-up care and Rehabilitation Geriatric.

The investigators assume that the application of a procedure based on osteopathic fascial techniques in elderly care in Suite and Geriatric Rehabilitation ( SSRG ) suffering from pain of nursing care, could reduce the painful phenomenon having systemic action, and improve tissue engineering, trophicity viscera and the neurovascular supply .

DETAILED DESCRIPTION:
The prevalence of pain in the elderly is very important, especially for people living in institutions ( 40-70 % according to recent studies). Among the most common complaints include pain induced by treatments. It is defined by Upsa Laboratory as pain of "short duration caused by the caregiver in the foreseeable occurrence of circumstances and can be prevented by suitable measures ." Responsible care are induced pain dressings, levies and other diagnostics actions, mobilizations during an exchange , a toilet, a transfer between different services or an act of rehabilitation. The repetition of acts and therefore the pain , is also a source of anxiety for older people who often have to anticipate the following treatments , and thus hinder the care relationship.

The evaluation of the induced pain is a growing concern for all caregivers. It concerns all the players care, medical or paramedical.

Prevention and relief of pain induced is part of regulatory obligations become since the Law of 4 March 2002 on patients' rights and quality of the health system. It is in this dynamic, in 2006 the Ministry of Health and Solidarity launched a support plan to improve the pain, one of whose objectives was to promote the quality of life of older people reducing the impact of pain on daily life.

To assess pain in seniors several scales are listed and validated: ECPA scale that allows the evaluation of recurrent pain induced pain and is used in some service of Suite and Geriatric Rehabilitation (SSRG); Doloplus scale is more suitable for evaluation of chronic pain and finally Algoplus scale specialized in the evaluation of acute pain. The pain assessment difficulties in the elderly are also accentuated by the many possible etiologies, the fatalistic attitude of some and the belief that pain is part of a normal aging process.

It is therefore to identify the intensity of the pain, its characteristics and causes to guide treatment. The pain relief will be based on non-drug means (prevention, care explanation, hypnosis, massage, cryotherapy), and / or medication when analgesia is no longer sufficient. Drug treatment, however, have the disadvantage of frequent side effects and be difficult to use in the elderly already poly medicated. Non-drug therapies, they can help limit the requirements, and therefore their side effects, and as such are to be considered in addition to usual care.

Osteopathy is a holistic manual medicine that aims to prevent and remedy various functional disorders of the body. This discipline has a wide scope whose positive influence was demonstrated on particular musculoskeletal pain type of neck pain, back pain, visceral on as chronic constipation, gastric reflux, migraines, or back pain chronic in the elderly in institutions.

This study's main objective is to determine through a randomized controlled clinical trial, the efficacy of osteopathy on the reduction of pain induced in the elderly in institutions.

This type of study can have an impact on public health policy and help improve :

* the treatment of pain induced in people SSRG ;
* propose a better use of medication and non-pharmacological methods like osteopathy ;
* assist in structuring the health care sector.

The public will be randomized using a block randomization, into two groups: a "osteopathy" group and a "simulated" group (simulated techniques).

Both procedures will not be provided by the same operator. Two exclusive osteopathic will load groups "osteopathy" and "simulated" according to randomization to be set so as to ensure a random distribution of the groups, that is to say, each operator will be as many patients that simulated .

Service nurses will be in charge of data collection, blind, that is to say that they have knowledge that the patient is included in the study but not the membership group. This methodology will allow us as well to justify the contribution of osteopathy in relation to the natural course of the patient's health status, and to justify the contribution of osteopathy regardless of the operator. Operators will support different patients included in the study in the same way, regardless of their allocation group. Thus, it will be applied a standardized osteopathic and simulated procedure (described above) and the same attitude of support from operators. Including verbal exchanges will be the same, addressing different areas of the patient, whether medical, family, or professional. The goal is to ensure some standardization in the management, which standardizes the simulated treatment and making it look like at any point in the care osteopathic. For the sake of continuity of treatment, it is "osteopathic" or "simulated" the operator assigned after randomization will perform the 3 sessions with the same patient.

-Group " osteopathy ": an osteopathic fascial only procedure will be used , having no technique called " impulsive " (or Thrust technique during which the patient may hear a cracking sound ) . This approach therefore does not present any particular risk of side effects for the patient.

Specifically , the following techniques will be applied by the operator in order that wish to: A technical on (or) scar (s)

* Technical overall equilibration of the upper limbs
* Technical overall equilibration of the lower limbs
* A basic technique spread
* Technical C0 of equilibration relative to the sternum
* A technique of diaphragmatic equilibration
* A fascial technique on dorsal vertebrae and / or lumbar

At protocol performed for osteopathy group will be assigned to each area addressed by each technique a coefficient of osteopathic dysfunction assessed in this way:

* Lack of dysfunction, coefficient 0
* low Dysfunction, coefficient equal to 1
* moderate dysfunction, coefficient equal to 2
* strong Dysfunction, coefficient equal to 3 These coefficients will be recorded in a table at each meeting and will allow the operator to monitor the patient own dysfunctional pattern.
* Group " simulated ": The simulated protocol similar to that used in the study of John C. Licciardone et al. and validated by North Texas Chronic Low Back Pain Trial , is performed in the same positions as the care osteopathic . The operator places his hands on the same areas , avoiding associated mobilize joints and muscles.

Both procedures " osteopathic " and "simulated" , will be provided in three sessions lasting 60 minutes each, one week apart . The interval of one week is justified by the fact that the nursing care can be repeated several times a day , and the constraints of prolonged bed rest being permanent , the tissues of patients are found in an advanced state of fibrosis . It then seems necessary to allow an integration time between sessions. The choice of 3 sessions is based on a compromise between feasibility in the service, acceptability for the patient and the investigators' assessment of the optimal intensity of the procedure. Week 4 , only a data collection will be realized.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 75 years ;
* Patients residing in Suite Care service and Geriatric Rehabilitation with pain induced by the nursing care;
* Pain intensity measured by the Behavioral Assessment Scale of pain in the Aged Person ( ECPA) at least 8/32 within five days before the start of the study;
* Patients having informed and signed a free and informed consent ;
* Affiliated to social security scheme (beneficiary or assignee ) .

Exclusion Criteria:

* Medical contraindication to the practice of osteopathy ;
* Osteopathic treatment during the past year ;
* Patients under tutorship and curatorship .

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Care-induced Pain assessed by Behavioural Scale | Every week after inclusion during 4 weeks
  Behavioural Scale to Evaluate Pain in Non-communicating Adults (ECPA)

SECONDARY OUTCOMES:
Evaluation of variation in the Consumption of Analgesics (frequency, dose, type) | Every day from inclusion during 4 weeks
  Consumption of analgesics will be measured with the name of drug, the frequency and the dose Measure : Comparison of analgesic consumption before and after 3 sessions of osteopathy ( between S0 and S4) : increase or decrease the frequency, dose or type
Evaluation of Pain | 4 weeks
  Visual Analog Scale (VAS) for communicating Adults or Algoplus Scale for non-communicating Adults

CONTACTS AND LOCATIONS:
Overall Officials: Martine MERCERON, PH, Principal Investigator — René Dubos Hospital (PONTOISE-FRANCE)
Locations (2):
- France (2):
  - Intercommunal Hospital Group of Vexin - Geriatric care and rehabilitation department, Marines
  - René Dubos Hospital - Geriatric care and rehabilitation department, Pontoise, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No